CLINICAL TRIAL: NCT00078156
Title: Women's Treatment for Trauma and Substance Use Disorders
Brief Title: Women's Treatment for Trauma and Substance Use Disorders - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Denise Hien, Ph.D., New York State Psychiatric Institute
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-CTN-0015-1
Record Dates: First submitted 2004-02-19; First posted 2004-02-23 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Substance-Related Disorders
Keywords: behavioral intervention
MeSH Terms: conditions — Substance-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to compare the effectiveness of adding Seeking Safety to standard substance abuse treatment to adding a control condition: Women's Health Education to standard substance abuse treatment.

ELIGIBILITY:
Inclusion Criteria - Women with a diagnosis of substance abuse or dependence who also have either full or sub-threshold DSM-IV PTSD.

Exclusion Criteria:

- Women will be excluded from the study who have current psychotic disorders, or a history of active psychosis (past two months); women with a diagnosis of substance abuse or dependence who also have either full or sub-threshold DSM-IV PTSD; and women who have current psychotic disorders, or a history of active psychosis (past two months).

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409
Dates: Start 2004-01; Primary Completion 2005-10 (Actual); Study Completion 2005-10

PRIMARY OUTCOMES:
Drug abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Denise Hien, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (7):
- United States (7):
  - Gateway Community Services, Jacksonville, Florida
  - The Villiage, Miami, Florida
  - Addiction Research & Treatment Corp.-MSUCAS, Brooklyn, New York
  - Addiction Research & Treatment Corp.-RISE, Brooklyn, New York
  - Maryhaven, Inc., Columbus, Ohio
  - Charleston Center, Charleston, South Carolina
  - Residence XII, Kirkland, Washington

REFERENCES:
- [Derived] Ruglass LM, Shevorykin A, Zhao Y, Killeen TK, Bauer AG, Morgan-Lopez AA, Back SE, Fitzpatrick S, Lopez-Castro T, Norman SB, Saavedra LM, Hien DA. Self-report and urine drug screen concordance among women with co-occurring PTSD and substance use disorders participating in a clinical trial: Impact of drug type and participant characteristics. Drug Alcohol Depend. 2023 Mar 1;244:109769. doi: 10.1016/j.drugalcdep.2023.109769. Epub 2023 Jan 14. PMID 36696843
- [Derived] Fitzpatrick SS, Morgan-Lopez AA, Saraiya TC, Back SE, Killeen TK, Norman SB, Lopez-Castro T, Ruglass LM, Saavedra LM, Hien DA. Graded response item response theory in scaling suicidal thoughts and behaviors among trauma-exposed women with substance use disorders. Psychol Addict Behav. 2022 Jun;36(4):397-409. doi: 10.1037/adb0000757. Epub 2021 Jun 17. PMID 34138594
- [Derived] Saavedra LM, Morgan-Lopez AA, Hien DA, Killeen TK, Back SE, Ruglass LM, Fitzpatrick S, Lopez-Castro T. Putting the Patient Back in Clinical Significance: Moderated Nonlinear Factor Analysis for Estimating Clinically Significant Change in Treatment for Posttraumatic Stress Disorder. J Trauma Stress. 2021 Apr;34(2):454-466. doi: 10.1002/jts.22624. Epub 2020 Nov 11. PMID 33175470
- [Derived] Ruglass LM, Morgan-Lopez AA, Saavedra LM, Hien DA, Fitzpatrick S, Killeen TK, Back SE, Lopez-Castro T. Measurement nonequivalence of the Clinician-Administered PTSD Scale by race/ethnicity: Implications for quantifying posttraumatic stress disorder severity. Psychol Assess. 2020 Nov;32(11):1015-1027. doi: 10.1037/pas0000943. Epub 2020 Aug 27. PMID 32853005
- [Derived] Morgan-Lopez AA, Killeen TK, Saavedra LM, Hien DA, Fitzpatrick S, Ruglass LM, Back SE. Crossover between diagnostic and empirical categorizations of full and subthreshold PTSD. J Affect Disord. 2020 Sep 1;274:832-840. doi: 10.1016/j.jad.2020.05.031. Epub 2020 May 24. PMID 32664022
- [Derived] Hameed M, O'Doherty L, Gilchrist G, Tirado-Munoz J, Taft A, Chondros P, Feder G, Tan M, Hegarty K. Psychological therapies for women who experience intimate partner violence. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013017. doi: 10.1002/14651858.CD013017.pub2. PMID 32608505
- [Derived] Morgan-Lopez AA, Saavedra LM, Hien DA, Killeen TK, Back SE, Ruglass LM, Fitzpatrick S, Lopez-Castro T, Patock-Peckham JA. Estimation of equable scale scores and treatment outcomes from patient- and clinician-reported PTSD measures using item response theory calibration. Psychol Assess. 2020 Apr;32(4):321-335. doi: 10.1037/pas0000789. Epub 2019 Dec 5. PMID 31804102
- [Derived] Resko SM, Brown S, Mendoza NS, Crosby S, Gonzalez-Prendes A. Perceived Treatment Needs Among Women With Co-occurring Substance Use Disorders and PTSD. J Dual Diagn. 2016 Jul-Dec;12(3-4):271-281. doi: 10.1080/15504263.2016.1248309. Epub 2016 Oct 14. PMID 27739935
- [Derived] Lopez-Castro T, Hu MC, Papini S, Ruglass LM, Hien DA. Pathways to change: Use trajectories following trauma-informed treatment of women with co-occurring post-traumatic stress disorder and substance use disorders. Drug Alcohol Rev. 2015 May;34(3):242-51. doi: 10.1111/dar.12230. Epub 2015 Mar 4. PMID 25735200
- [Derived] Morgan-Lopez AA, Saavedra LM, Hien DA, Campbell AN, Wu E, Ruglass L, Patock-Peckham JA, Bainter SC. Indirect effects of 12-session seeking safety on substance use outcomes: overall and attendance class-specific effects. Am J Addict. 2014 May-Jun;23(3):218-25. doi: 10.1111/j.1521-0391.2014.12100.x. PMID 24724878
- [Derived] Ruglass LM, Hien DA, Hu MC, Campbell AN. Associations between post-traumatic stress symptoms, stimulant use, and treatment outcomes: a secondary analysis of NIDA's Women and Trauma study. Am J Addict. 2014 Jan-Feb;23(1):90-5. doi: 10.1111/j.1521-0391.2013.12068.x. Epub 2013 Jun 26. PMID 24313246
- [Derived] Morgan-Lopez AA, Saavedra LM, Hien DA, Campbell AN, Wu E, Ruglass L. Synergy between seeking safety and twelve-step affiliation on substance use outcomes for women. J Subst Abuse Treat. 2013 Aug;45(2):179-89. doi: 10.1016/j.jsat.2013.01.015. Epub 2013 Apr 1. PMID 23558158
- [Derived] Hien DA, Morgan-Lopez AA, Campbell AN, Saavedra LM, Wu E, Cohen L, Ruglass L, Nunes EV. Attendance and substance use outcomes for the Seeking Safety program: sometimes less is more. J Consult Clin Psychol. 2012 Feb;80(1):29-42. doi: 10.1037/a0026361. Epub 2011 Dec 19. PMID 22182262
- [Derived] Hien DA, Jiang H, Campbell AN, Hu MC, Miele GM, Cohen LR, Brigham GS, Capstick C, Kulaga A, Robinson J, Suarez-Morales L, Nunes EV. Do treatment improvements in PTSD severity affect substance use outcomes? A secondary analysis from a randomized clinical trial in NIDA's Clinical Trials Network. Am J Psychiatry. 2010 Jan;167(1):95-101. doi: 10.1176/appi.ajp.2009.09091261. Epub 2009 Nov 16. PMID 19917596
- [Derived] Hien DA, Wells EA, Jiang H, Suarez-Morales L, Campbell AN, Cohen LR, Miele GM, Killeen T, Brigham GS, Zhang Y, Hansen C, Hodgkins C, Hatch-Maillette M, Brown C, Kulaga A, Kristman-Valente A, Chu M, Sage R, Robinson JA, Liu D, Nunes EV. Multisite randomized trial of behavioral interventions for women with co-occurring PTSD and substance use disorders. J Consult Clin Psychol. 2009 Aug;77(4):607-19. doi: 10.1037/a0016227. PMID 19634955
- [Derived] Hien DA, Campbell AN, Killeen T, Hu MC, Hansen C, Jiang H, Hatch-Maillette M, Miele GM, Cohen LR, Gan W, Resko SM, DiBono M, Wells EA, Nunes EV. The impact of trauma-focused group therapy upon HIV sexual risk behaviors in the NIDA Clinical Trials Network "Women and trauma" multi-site study. AIDS Behav. 2010 Apr;14(2):421-30. doi: 10.1007/s10461-009-9573-7. Epub 2009 May 19. PMID 19452271